CLINICAL TRIAL: NCT03479385
Title: Developing an Integrative Intervention for Breast Cancer Survivorship
Brief Title: Integrative Approaches to Cancer Survivorship: Project 3
Acronym: IACS2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 16-185671
Record Dates: First submitted 2018-03-20; First posted 2018-03-27 (Actual); Last update posted 2020-03-25 (Actual); Status verified 2020-03

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Integrative Medicine Intervention (Experimental): Study participants randomized to the Integrative Medicine intervention will attend 14 sessions with an Integrative Medicine clinician over the course of 6 months potentially followed by a 6 month maintenance phase. The treatment modalities employed in the study will include nutrition and lifestyle recommendations.
  Interventions: Behavioral: Integrative Medicine Intervention
- Health Education Intervention (Experimental): Study participants randomized to the Health Education intervention will attend 14 sessions with a Health Educator over the course of 6 months. The emphasis in the sessions will be to provide engaging educational information on common survivorship issues.
  Interventions: Behavioral: Health Education Intervention

INTERVENTIONS:
Behavioral: Integrative Medicine Intervention — Study participants will attend 14 sessions with an Integrative Medicine clinician over the course of 6 months, potentially followed by a 6 month maintenance phase.
  Arms: Integrative Medicine Intervention
Behavioral: Health Education Intervention — Study participants will attend 14 sessions with a Health Educator over the course of 6 months.
  Arms: Health Education Intervention

SUMMARY:
The purpose of this study is to conduct a randomized controlled trial or RCT of the following 2 supportive care interventions in recent breast cancer survivors: an Integrative Medicine intervention based on Ayurvedic medicine and a Health Education intervention.

DETAILED DESCRIPTION:
Post-treatment cancer survivorship is often associated with a void in care given the drop-off in support provided to survivors from the medical team as well as family and friends. In addition, cancer associated symptoms and impaired quality of life remain significant problems for patients despite advances in cancer treatment. Few effective treatment options exist for these symptoms. Integrative medicine is rising in popularity in the United States; however, few integrative medicine modalities have been rigorously studied. Ayurveda, a whole system of medicine that originated in the Indian subcontinent, has its own system of diagnostics and therapeutics, and among its strengths are wellness and prevention. In the Integrative Medicine intervention, Ayurvedic nutrition and lifestyle guidance will be presented, along with instruction in Yoga. In the Health Education intervention, informative content on issues relevant to breast cancer survivors will be presented including the physical, social and emotional impacts of survivorship. The investigators aim to perform a pilot RCT in breast cancer survivors with impaired quality of life. Specifically, the investigators aim to assess feasibility of randomization, adherence and retention to the Integrative Medicine and Health Education interventions.

ELIGIBILITY:
Inclusion Criteria:

* Female breast cancer survivor who is over 1 month and less than 24 months beyond the completion of primary therapy (surgery, radiation, and chemotherapy)
* Having received chemotherapy as part of their primary therapy for breast cancer
* Be in complete remission
* Aged 18 years or older
* Able to read, write, and understand English
* Karnofsky Performance Status (KPS) greater than or equal to 60
* Have impaired quality of life
* Ability to give informed consent

Exclusion Criteria:

* Having received Ayurvedic treatment within 6 months of study enrollment
* Receiving chemotherapy or radiotherapy at the time of study enrollment. Anti-her2 directed therapy is not exclusionary.
* Being within 1 month (before or after) of surgery for breast cancer (including breast reconstructive surgery). Smaller surgical procedures such as implant exchange are not exclusionary.
* Patients on adjuvant hormone therapy for less than 2 months
* Have surgery for breast cancer or breast reconstructive surgery planned during the initial 6 month study period. Smaller surgical procedures such as implant exchange are not exclusionary.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-04-17 (Actual); Primary Completion 2019-02-06 (Actual); Study Completion 2020-01-30 (Actual)

PRIMARY OUTCOMES:
Change in quality of life over 6 months | Baseline, 3 months, 6 months
  The investigators will use the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ C30) in conjunction with a breast cancer-specific subscale, BR23, to collect data on qualify of life and cancer-related symptoms.
  The scales range in score from 0 to 100. A high scale score represents a higher response level. Thus a high score for a functional scale represents a high / healthy level of functioning, a high score for the global health status / QoL represents a high QoL, but a high score for a symptom scale / item represents a high level of symptomatology / problems.
  The principle for scoring these scales is the same in all cases:
  1. Estimate the average of the items that contribute to the scale; this is the raw score.
  2. Use a linear transformation to standardise the raw score, so that scores range from 0 to 100; a higher score represents a higher ("better") level of functioning, or a higher ("worse") level of symptoms.

SECONDARY OUTCOMES:
Change in fatigue over 6 months | Baseline, 3 months, 6 months
  The investigators will use the Lee Fatigue Scale (LFS) to collect data on fatigue.
  The scale ranges from 0 - 10. Scoring Instructions: To interpret it clinically, it is good to think about the lower 1/3 scores (0-3.2) being none or minimal fatigue, the middle 1/3 (3.3 to 6.6) being moderate fatigue, and the top 1/3 (6.7 to 10) being high fatigue.
  * Energy Item Score: Mean of items 6-10
  * Fatigue Item Score: Mean of 1-5 and 11-18
Change in sleep quality over 6 months | Baseline, 3 months, 6 months
  The investigators will use the General Sleep Disturbance Scale (GSDS) to collect data on sleep disturbance.
  The scale ranges from 0 (never) - 7 (Every Day) Reverse score items: 4, 10, 11, 12 (e.g., 0=7, 1=6, 2=5, 3=4, 4=3, 5=2, 6=1, 7=0).
  Scoring Instructions:
  * Total Sum Score (gstot): Mean of all items * 21 (must have at least 16 items scored)
  * Medications for Sleep Sum Score (gsmed): Mean of items 16-21 * 16 (must have at least 4)
  * Quality of Sleep Sum Score (gsqal): Mean of items 4, 5, 10 * 3 (must have at least 2)
  * Quantity of Sleep Sum Score (gsqnt): Mean of items 12, 13 * 2 (must have at least 2)
  * Sleep Onset Latency (gsol): Item 1
  * Mid Sleep Wakes (gsmid): Item 2
  * Early Awakenings (gsend): Item 3
  * Excessive Daytime Sleepiness Sum Score (gseds): Mean of 6, 7, 8, 9, 11, 14, 15 * 7 (must have at least 5)
Change in anxiety over 6 months | Baseline, 3 months, 6 months
  The investigators will use the Spielberger State Anxiety Inventory (STAI-S) to collect data on anxiety.
  The scale ranges from 1 (Not at all) - 4 (Very much so) Reverse Scoring Items: 1, 2, 5, 8, 10, 11, 15, 16, 19, 20 Outcome Variables: Scores range between 20-80
  * Total Sum Score (no missing values): Sum all questions
  * Total Sum Score (few items missing): Average of the non-missing items and multiply by 20.
Change in depressive symptoms over 6 months | Baseline, 3 months, 6 months
  The investigators will use the Center for Epidemiological Studies - Depression Scale (CES-D) to collect data on depressive symptoms.
  The scale ranges from 0 (Rarely) - 3 (Most Days) Reverse Scoring Items: 4, 8, 12, 16 Outcome Variables: Scores range between 0-60. If participant scores higher than 16, refer to guidelines for CES-D
  • Total Sum Score: Sum of 20 questions. Do not score if more than 4 missing answers.
Change in pain over 6 months | Baseline, 3 months, 6 months
  The investigators will use the Brief Pain Inventory (BPI) to collect data on pain intensity and interference with function.
Change in diet over 6 months | Baseline, 3 months, 6 months
  The investigators will use the Automated Self-Administered 24-hour Recall (ASA24) to assess dietary recall over a 24 hour period.

CONTACTS AND LOCATIONS:
Overall Officials: Anand Dhruva, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, Osher Center for Integrative Medicine, San Francisco, California, United States